CLINICAL TRIAL: NCT06446245
Title: DIRECT: Doxycycline Adjunctive Therapy to Reduce Excess Mortality and Complications From Central Nervous System Tuberculosis - Phase II Randomized Clinical Trial
Brief Title: Adjunctive Doxycycline for Central Nervous System Tuberculosis
Acronym: DIRECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024/00039
Record Dates: First submitted 2024-05-28; First posted 2024-06-06 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis, Meningeal; Tuberculosis; Meningitis (Etiology); Tuberculosis, Central Nervous System; Tuberculosis; Meningoencephalitis (Etiology)
MeSH Terms: conditions — Tuberculosis, Meningeal; Tuberculosis; Meningitis; Tuberculosis, Central Nervous System; Meningoencephalitis | interventions — Doxycycline; Antitubercular Agents

STUDY DESIGN:
Intervention Model Description: Phase II, multi-center randomised controlled trial, parallel design of intervention versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline + standard anti-tuberculous treatment + corticosteroid therapy (Experimental): Doxycycline 100 mg twice daily with once daily anti-tuberculous treatment comprising of at least three agents, including rifampicin 10 mg/kg, isoniazid 5 mg/kg, ethambutol 15 - 20 mg/kg, ± pyrazinamide 25 mg/kg and pyridoxine 10-50 mg per day, or aminoglycosides or quinolones according to managing physicians' discretion. Adjunctive corticosteroids to be dosed at 0.4mg/kg/day of dexamethasone or equivalent for week 1, then 0.3mg/kg/day for week 2, 0.2mg/kg/day for week 3, 0.1mg/kg/day for week 4, then tapered to stop over the next 4 weeks. Other forms of corticosteroids are also acceptable e.g. hydrocortisone, methylprednisolone at the equivalent dosage. Where needed, the drugs will be adjusted according to renal function. These will be given daily for 8 weeks. Subsequently doxycycline will be ceased and patients are to continue with their standard anti-tuberculous treatment and duration according to their managing physician.
  Interventions: Drug: Doxycycline; Drug: Anti Tuberculosis Drug; Drug: Adjunctive corticosteroid
- Placebo + standard anti-tuberculous treatment + corticosteroid therapy (Placebo Comparator): Placebo twice daily with once daily anti-tuberculous treatment comprising of at least three agents, including rifampicin 10 mg/kg, isoniazid 5 mg/kg, ethambutol 15-20 mg/kg, ± pyrazinamide 25 mg/kg and pyridoxine 10-50 mg per day, or aminoglycosides or quinolones according to managing physicians' discretion. Adjunctive corticosteroids to be dosed at 0.4mg/kg/day of dexamethasone or equivalent for week 1, then 0.3mg/kg/day for week 2, 0.2mg/kg/day for week 3, 0.1mg/kg/day for week 4, then tapered to stop over the next 4 weeks. Other forms of corticosteroids are also acceptable e.g. hydrocortisone, methylprednisolone at the equivalent dosage. Where needed, the drugs will be adjusted according to renal function. These will be given daily for 8 weeks. Subsequently placebo will be ceased and patients are to continue with their standard anti-tuberculous treatment and duration according to their managing physician.
  Interventions: Drug: Placebo; Drug: Anti Tuberculosis Drug; Drug: Adjunctive corticosteroid

INTERVENTIONS:
Drug: Doxycycline — adjunctive doxycycline to standard anti-tuberculous treatment and corticosteroid therapy
  Arms: Doxycycline + standard anti-tuberculous treatment + corticosteroid therapy
Drug: Placebo — Placebo
  Arms: Placebo + standard anti-tuberculous treatment + corticosteroid therapy
Drug: Anti Tuberculosis Drug — Standard anti-tuberculous therapy
Drug: Adjunctive corticosteroid — Adjunctive corticosteroids to be dosed at 0.4mg/kg/day of dexamethasone or equivalent for week 1, then 0.3mg/kg/day for week 2, 0.2mg/kg/day for week 3, 0.1mg/kg/day for week 4, then tapered to stop over the next 4 weeks. Other forms of corticosteroids are also acceptable eg. hydrocortisone, methylprednisolone at the equivalent dosage

SUMMARY:
Although tuberculosis is now considered a treatable disease, central nervous system tuberculosis (CNS-TB) when managed with the current standard-of-care (SOC), still has mortality rates ranging from 30-50% even in tertiary hospital centers. At present, the SOC for the management of CNS-TB is anti-tuberculous therapy with adjunctive corticosteroids. In CNS-TB, the activity of pathogenic host matrix metalloproteinases (MMPs) is unopposed to tissue inhibitors of metalloproteinases (TIMPs), resulting in a matrix-degrading phenotype which may drive worse outcomes in CNS-TB. In a prior established CNS-TB murine model, the investigators have demonstrated that adjunctive MMP inhibition using doxycycline, a widely available and cheap drug, in addition to standard TB treatment, compared with standard TB treatment alone, improved murine survival (Manuscript in preparation). The investigators previously showed that in humans with pulmonary TB, doxycycline with anti-TB treatment is safe, accelerates the resolution of inflammation, and suppresses systemic and respiratory MMPs. Hence, the investigators are now ideally positioned to determine if adjunctive doxycycline in patients with CNS-TB can improve clinical outcomes. The investigators will perform a Phase 2 double-blind randomized-controlled trial (RCT) of adjunctive doxycycline versus placebo with standard TB treatment and steroids for 8 weeks, with the primary outcome of 8-week mortality or severe neurological deficits.

DETAILED DESCRIPTION:
The investigators hypothesize that in patients with CNS-TB, the addition of doxycycline to SOC improves clinical outcomes.

The specific aims are to determine:

1. Whether the primary outcome of mortality rates or severe neurological deficits in CNS-TB patients in the doxycycline arm improves at 8 weeks. Neurological deficits will be defined using a modified Rankin scale score of 3 or higher to measure the degree of disability or dependence in the daily activities of people who have suffered from neurological disability.
2. Whether MMPs and inflammatory gene transcriptomics in the doxycycline arm are reduced. Plasma and cerebrospinal fluid (CSF) MMPs and TIMPs will be measured by luminex bead array technology. The functional activity of CSF MMPs will be assessed using Dye-quenched (DQ) Gelatin degradation. Inflammatory gene transcripts will be measured using whole-blood bulk RNA sequencing and single-cell RNA sequencing. CSF will also be profiled using single-cell RNA sequencing.
3. Whether concurrent SOC treatment and doxycycline for CNS-TB are safe. The investigators will monitor patients for side effects including liver function tests to evaluate any significant change in the safety profile of the patients after administration of adjunctive doxycycline, in comparison to the placebo arm. Standard measures such as grade 3 or 4 adverse events or serious adverse events will be determined.

These specific aims will determine if doxycycline will improve clinical outcomes in the management of CNS-TB, reduce long-term neurological deficits whilst demonstrating a comparable safety profile. These aims are critical to form the basis of a large-scale Phase 3 randomised-controlled trial of CNS-TB which will positively impact clinical practice and international guidelines.

Background and Clinical Significance

The global burden of tuberculosis and TB sequelae

Despite being declared an emergency by the World Health Organisation (WHO) in 1993, tuberculosis (TB) remains a global health epidemic. A significant proportion of the global population is infected with TB, particularly in lower- to middle-income countries in resource-limited settings. Despite strategies directed towards infection control and TB management, worldwide annual TB deaths are estimated to be 1.3 million. Furthermore, the coronavirus disease 2019 (COVID-19) pandemic has also impacted TB, and TB incidence is expected to rise substantially. In Singapore, TB incidence has stagnated after some significant improvements with an annual incidence of approximately 39 TB infections per 100,000 people, which translates to under 3,000 TB patients per year. Additionally, there are rising multi-drug-resistant (MDR) and extensively drug-resistant (XDR) TB regionally and in the world, which pose clinical challenges. MDR and XDR TB often require prolonged treatment courses with medications that are often unavailable in resource-limited settings. Singapore is not exempted from the scourge of MDR and XDR TB cases, which have been described in prisons, gaming arcades and even housing estates. Global and local epidemiology indicates that TB remains an infectious disease threat.

One of the most severe forms of TB is CNS-TB which can lead to significant morbidity and mortality. In CNS-TB, tissue destruction can result in long-term neurological sequelae with permanent neurological deficits. Even with appropriate treatment for CNS-TB and microbiological cure, mortality rates for CNS-TB remain high at up to 30-50%; CNS-TB may still leave behind residual neurological deficits. Patients can become bed-bound and dependent on activities of daily living. Even with good standard-of-care, there still is cognitive impairment in up to 55% of patients and motor deficits in up to 40% of patients, with significant residual neurological deficits. Adjunctive steroids significantly reduce mortality (41.3% placebo vs 31.8% in the steroid arm), but death rates remain unacceptably high. Critically, steroids did not show a significant improvement in severe disability from neurological deficits. TB sequelae cause substantial morbidity long after TB itself is treated, as currently there is no treatment to prevent severe neurological disability.

Host immunopathology and TB tissue destruction

Prior published work has shown that the cause of tissue destruction in TB resulting in sequelae is excessive host inflammatory and adaptive immune response. Although the immunopathology in TB is not fully understood, it has been shown that pro-inflammatory cytokines such as tumour necrosis factor-alpha (TNF-α) may play a key role. Proteases result in tissue destruction in TB patients, with MMPs having a unique ability to collectively degrade all extracellular matrix fibrils at a neutral power of hydrogen (pH), of which the secretion of MMPs in TB is excessive. MMP activity is dysregulated in TB, which is the key in the pathophysiology. The secretion of multiple MMPs are up-regulated, arising from human macrophages, epithelial cells and neutrophils which we showed. The upregulation of MMPs with tissue destruction has been shown in several TB animal models, which provides further evidence on the role of pathogenic MMPs in vivo.

Doxycycline is the only MMP inhibitor licensed by the U.S. Food and Drug Administration which has both anti-bacterial and immunomodulatory properties. It is an antibiotic that is used for decades for a range of clinical indications, including periodontal disease (gum disease), acting on periodontal clefts by reducing the concentration of collagenases. Doxycycline has also been shown to be bacteriostatic to Mycobacterium tuberculosis (Mtb). It has an excellent safety profile, even when given for prolonged durations. It may also be administered by nasogastric tube for individuals with swallowing disability. Furthermore, it is a drug that is widely available and cheap, making it highly accessible even in resource-limited settings. The addition of doxycycline adjunctive therapy to corticosteroids and standard TB therapy may decrease host MMP expression and inflammatory gene responses in human CNS-TB, hence improving clinical outcomes and neurological sequelae.

Doxycycline modulates TB tissue destruction

The first doxycycline pulmonary TB trial worldwide was conducted by us. In a Phase 2 double-blind randomised-controlled trial of 30 pulmonary TB patients, investigating doxycycline host-directed therapy funded by the National Medical Research Council, the investigators showed that 2 weeks of doxycycline improved pulmonary cavity resolution as indicated by the patients exhibiting significantly smaller cavities. In addition, there was also a beneficial host immunological effect that persisted 6 weeks post-discontinuation of the doxycycline, accelerating a return to healthy gene expression of the host transcriptome. MMPs were also down-regulated with suppression of plasma MMP-1 and further reduction of collagenase and gelatinase MMPs in the sputum. However, the effects of doxycycline on mortality or neurological outcomes in CNS-TB are unknown. This Phase 2 randomised-controlled-trial determines if adjunctive doxycycline treatment can be extended to CNS-TB to improve clinical outcomes and neurological sequelae. Reducing neurological disability would alleviate burden on healthcare facilities and maximise an individual's economically productive life. If positive, these findings will provide preliminary data for a Phase 3 RCT. Findings will be rapidly conveyed to the WHO with whom the investigators closely collaborate, to impact international guidelines and clinical practice.

Specific Aims and Hypothesis

The investigators hypothesize that in patients with CNS-TB, the addition of doxycycline to SOC improves clinical outcomes.

The specific aims are to determine:

1. Whether the primary outcome of mortality rates or severe neurological deficits in CNS-TB patients in the doxycycline arm improves at 8 weeks. Neurological deficits will be defined using a modified Rankin scale score of 3 or higher to measure the degree of disability or dependence in the daily activities of people who have suffered from neurological disability.
2. Whether MMPs and inflammatory gene transcriptomics in the doxycycline arm are reduced. Plasma and cerebrospinal fluid (CSF) MMPs and TIMPs will be measured by luminex bead array technology. The functional activity of CSF MMPs will be assessed using Dye-quenched (DQ) Gelatin degradation. Inflammatory gene transcripts will be measured using whole-blood bulk RNA sequencing and single-cell RNA sequencing. CSF will also be profiled using single-cell RNA sequencing.
3. Whether concurrent SOC treatment and doxycycline for CNS-TB are safe. The investigators will monitor patients for side effects including liver function tests to evaluate any significant change in the safety profile of the patients after administration of adjunctive doxycycline, in comparison to the placebo arm. Standard measures such as grade 3 or 4 adverse events or serious adverse events will be determined.

These specific aims will determine if doxycycline will improve clinical outcomes in the management of CNS-TB, reduce long-term neurological deficits whilst demonstrating a comparable safety profile. These aims are critical to form the basis of a large-scale Phase 3 randomised-controlled trial of CNS-TB which will positively impact clinical practice and international guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 years and above.
2. Patients receiving ≤ 7 days of TB treatment or about to start combination TB treatment, including injectable agents, where required.
3. Patients with clinical evidence of TB meningitis, as per established diagnostic criteria, defined as either definite, probable or possible CNS-TB:

   1. "Definite" CNS-TB would be defined if acid-fast bacilli (AFB) or a positive nucleic acid amplification test for M. tuberculosis in the cerebrospinal fluid of patients.
   2. "Probable" CNS-TB would be defined if the patient exhibit one or more of the following: suspected pulmonary tuberculosis on chest radiography, acid-fast bacilli found in any specimen other than the cerebrospinal fluid or clinical evidence of other extrapulmonary tuberculosis.
   3. "Possible" CNS-TB would be defined if the patients exhibit at least four of the following: a history of tuberculosis, predominance of lymphocytes in the cerebrospinal fluid, a duration of illness of more than five days, a ratio of cerebrospinal fluid glucose to plasma glucose of less than 0.5, altered consciousness, yellow cerebrospinal fluid, or focal neurologic signs.
4. Alanine aminotransferase (ALT) level < 3 times the upper limit of normal.
5. Able to provide informed consent. If the patient has no mental capacity to give consent, then consent may be provided for by the patient's next of kin.
6. Lumbar puncture and brain imaging (either computed tomography or magnetic resonance imaging, with or without contrast) is required at baseline for enrolment

Exclusion Criteria:

1. Active Cancer
2. Pregnant or breastfeeding
3. Allergies to tetracyclines
4. Patients on retinoic acid, neuromuscular blocking agents or pimozide which may increase the risk of drug toxicity.
5. Autoimmune disease and/or on systemic immunosuppressants.
6. Use of any investigational or non-registered drug, vaccine or medical device other than the study drug within 182 days preceding dosing of the study drug or planned use during the study period.
7. Enrolment in any other clinical trial involving a systemic drug or intervention involving the CNS.
8. Contraindications to the use of steroids.
9. Investigators' assessment of lack of willingness to participate and comply with all requirements including follow-up of the protocol or identification of any factor presumed to significantly increase the participant's risk of suffering an adverse outcome.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mortality or severe neurological deficits (modified Rankin scale of 3 or more) at 8 weeks, from time of randomization. | 8 weeks
  Patients who survived at 8 weeks, from time of randomization, OR Persistent neurological disability at 8 weeks, from time of randomization, defined as a modified Rankin score of 3 or greater.

SECONDARY OUTCOMES:
Mortality at 8 weeks, from time of randomization | 8 weeks
  Mortality at 8 weeks, from time of randomization
Persistent neurological disability at 8 weeks, from time of randomization | 8 weeks
  Persistent neurological disability at 8 weeks, from time of randomization
Magnetic resonance imaging or Computed tomography brain at 8 weeks, from time of randomization, showing persistent changes associated with CNS-TB at 8 weeks, from time of randomization | 8 weeks
  Magnetic resonance imaging or Computed tomography brain at 8 weeks from time of randomization, showing persistent changes associated with CNS-TB, at 8 weeks, from time of randomization
The pattern of change of host transcriptome at week 8 from time of randomization | 8 weeks
  Whole blood will be collected in Tempus tubes and processed in a biosafety level-3 laboratory. Library preparation and bulk RNA sequencing will be performed as previously described. In addition, in the subset of patients recruited from Singapore, single-cell RNA sequencing (scRNAseq) will be performed from the doxycycline and placebo arm, analysing 10,000 cells per sample. In this subset of patients, blood for bulk RNAseq will also be stored as a backup. Single-cell RNAsequencing from the CSF will also be performed. Bioinformatic analyses will be performed to evaluate the pattern of change of host transcriptome at week 8, in established pipelines.
The pattern of change of host plasma MMPs at week 8 from time of randomization | 8 weeks
  Whole blood will be spun down, plasma collected and sterile filtered in a biosafety level-3 laboratory before transferring to a biosafety level-2 laboratory. MMP Luminex bead array will be performed which has been established in Dr Catherine Ong's laboratory. The pattern of change of host plasma MMPs at week 8.
The pattern of change of host CSF MMPs at week 2 from time of randomization | 2 weeks
  CSF will be collected and sterile filtered in a biosafety level-3 laboratory before transferring to a biosafety level-2 laboratory. MMP Luminex bead array will be performed which has been established in Dr Catherine Ong's laboratory. The host CSF MMPs at week 2 shall be evaluated.
Adverse events and serious adverse events | 8 weeks
  These will be recorded using the Division of AIDS table for Grading the Severity of Adult and Paediatric adverse events (December 2004)

CONTACTS AND LOCATIONS:
Locations (5):
- Indonesia (2):
  - Adam Malik Hospital, Medan
  - Universitas Sumatera Utara, Medan
- Sarawak General Hospital, Kuching, Sarawak, Malaysia
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Data may be made available on reasonable request

REFERENCES:
- [Background] Ong CW, Elkington PT, Friedland JS. Tuberculosis, pulmonary cavitation, and matrix metalloproteinases. Am J Respir Crit Care Med. 2014 Jul 1;190(1):9-18. doi: 10.1164/rccm.201311-2106PP. PMID 24713029
- [Background] Poh XY, Hong JM, Bai C, Miow QH, Thong PM, Wang Y, Rajarethinam R, Ding CSL, Ong CWM. Nos2-/- mice infected with M. tuberculosis develop neurobehavioral changes and immunopathology mimicking human central nervous system tuberculosis. J Neuroinflammation. 2022 Jan 24;19(1):21. doi: 10.1186/s12974-022-02387-0. PMID 35073927
- [Background] Miow QH, Vallejo AF, Wang Y, Hong JM, Bai C, Teo FS, Wang AD, Loh HR, Tan TZ, Ding Y, She HW, Gan SH, Paton NI, Lum J, Tay A, Chee CB, Tambyah PA, Polak ME, Wang YT, Singhal A, Elkington PT, Friedland JS, Ong CW. Doxycycline host-directed therapy in human pulmonary tuberculosis. J Clin Invest. 2021 Aug 2;131(15):e141895. doi: 10.1172/JCI141895. PMID 34128838